CLINICAL TRIAL: NCT06600776
Title: A Pilot Study Comparing the Efficacy of Dosing Ultra Rapid Insulin Lispro in a Medtronic 780G Hybrid Closed Loop System At Mealtime or Postmeal
Brief Title: Mealtime or Post-meal Dosing of URLi in Medtronic 780G Hybrid Closed Loop System
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLV-0332-24
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: Automated Insulin Delivery; Continuous Glucose Monitoring (CGM); Glycemic Control; Hybrid Closed Loop System; Insulin Bolus; Lyumjev; Mealtime Dosing; Medtronic 780G; Patient Preferences; Postmeal Dosing; Postprandial Glycemia; Time in Range (TIR); Type 1 Diabetes Mellitus (T1DM); Ultra Rapid Lispro Insulin (URLi)
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Patient Preference | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Intervention Model Description: Single Intervention Group: The study involves a single group of participants, all of whom are individuals with Type 1 Diabetes Mellitus (T1DM) using the Medtronic 780G hybrid closed-loop system with Ultra Rapid Lispro Insulin (URLi).
  Comparison Within Subjects: Participants will be asked to use the insulin dosing at mealtime during one period and post-meal during another. The study aims to compare the effects of premeal vs. post-meal dosing on glycemic control within the same group of individuals rather than comparing two different groups of participants.
  So, participants serve as their own control(in this case, mealtime vs. post-meal dosing).
Masking Description: Both the researchers and the participants are aware of the intervention being administered (premeal vs. post-meal dosing of Ultra Rapid Lispro Insulin). There is no blinding in the study, as participants will know when they are administering the insulin (whether at mealtime or post-meal), and the researchers will also have access to this information during data collection and analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Mealtime and Postmeal Dosing of Ultra Rapid Lispro Insulin (URLi) (Experimental): This arm consists of participants with Type 1 Diabetes Mellitus (T1DM) who are using the Medtronic 780G hybrid closed-loop system with Ultra Rapid Lispro Insulin (URLi). Participants will undergo two intervention phases: in one phase, URLi will be administered at mealtime (premeal dosing), and in the other phase, URLi will be administered immediately after meals (postmeal dosing). The dosage form is subcutaneous insulin infusion, and the insulin dose is based on individual carbohydrate counting. Each intervention phase will last for up to 4 weeks, with glycemic control and patient preferences assessed at the end of each phase.
  Interventions: Drug: Ultra Rapid Lispro (URLi); Device: Insulin pump with continuous glucose monitoring (CGM)

INTERVENTIONS:
Drug: Ultra Rapid Lispro (URLi) — Dosage Form:
  Subcutaneous insulin infusion
  Dosage:
  Based on individual carbohydrate counting, adjusted using the MiniMed 780G hybrid closed-loop system.
  Frequency:
  Administered at mealtime (premeal) during one phase and immediately after meals (postmeal) during the other phase.
  Duration:
  Each intervention phase lasts up to 4 weeks.
  Arm or Group/Intervention Cross-Reference:
  Both interventions (mealtime and postmeal dosing) are applied to the single arm of the study.
  Other Names: Lyumjev
Device: Insulin pump with continuous glucose monitoring (CGM) — The insulin pump with continuous glucose monitoring (CGM) system is used by patients with Type 1 Diabetes Mellitus (T1DM) as part of their regular treatment regimen. This system combines an insulin pump with real-time glucose monitoring, adjusting basal insulin delivery every 5 minutes based on continuous glucose data. In this study, participants are already using the system before the trial begins. The research does not examine the effect of the CGM itself but rather focuses on the timing of insulin bolus delivery (mealtime vs. postmeal) using their existing treatment system.
  Frequency:
  The system delivers basal insulin continuously and requires the patient to manually deliver bolus doses at mealtime (premeal) or postmeal, depending on the study phase.
  Duration:
  The device is used continuously throughout the entire study period, with each intervention phase (premeal vs. postmeal dosing) lasting up to 4 weeks.
  Arm or Group/Intervention Cross-Reference:
  This device will be us
  Other Names: MiniMed 780G Hybrid Closed-Loop System

SUMMARY:
This is a pilot study to compare premeal to postmeal dosing of ultra rapid lispro insulin (URLi) used in a MiniMed 780G system hybrid closed loop system. Subjects with type 1 diabetes mellitus (T1DM) already using a 780G hybrid closed loop system with URLi will be included. After signing a remote digital informed consent, a baseline record of the MiniMed 780G system will be downloaded from the Medtronic digital platform (Carelink system [1]) and subjects will be asked to fill an online questionnaire regarding their time of insulin dosing preferences and a 3-day online food diary [2]. During the intervention period subjects will be asked to provide a bolus dose of insulin only at the end of meals for up to 4 weeks. During the last week of the intervention period, subjects will be asked to fill out a 3-day online food diary [2]. At the end of the intervention period- a Carelink report [1] will be collected remotely and subjects will be asked to fill again the online questionnaire regarding their time of dosing preferences.

1. Primary Objective: To assess the efficacy of premeal dosing to post-meal dosing on parameters of glycemic control as obtained from continuous glucose monitoring.
2. Secondary Objective: To assess patient dosing preferences and the effect of premeal dosing vs. post-meal dosing on patient reported outcomes

Ref:

1. carelink.medtronic.eu
2. NutRatio.com.

ELIGIBILITY:
Inclusion Criteria:

Participants must be 18 years of age or older (inclusive).

Diagnosed with Type 1 Diabetes Mellitus (T1DM).

Already using the MiniMed 780G hybrid closed-loop system with Ultra Rapid Lispro Insulin (URLi) for at least 2 months prior to study enrollment.

Able and willing to provide informed consent electronically.

Willing and able to comply with the scheduled visits and other study procedures, including remote monitoring and completing questionnaires.

Exclusion Criteria:

Participants with a medical history of untreated active proliferative retinopathy.

Note: Subjects with non-proliferative retinopathy may be included. Subjects with treated proliferative retinopathy may be included based on the investigator's clinical judgment.

Severe acute or chronic medical or psychiatric conditions or laboratory abnormalities that may increase the risk associated with study participation or interfere with the interpretation of study results, as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-06 (Estimated); Primary Completion 2025-09-21 (Estimated); Study Completion 2025-10-21 (Estimated)

PRIMARY OUTCOMES:
Percentage of Time in Glucose Range (70-180 mg/dL) | Baseline to 4 weeks post-intervention
  The primary outcome measure is the percentage of time that blood glucose levels are within the target range of 70-180 mg/dL (Time in Range, TIR) as measured by continuous glucose monitoring (CGM). This will be compared between the mealtime dosing and postmeal dosing phases of Ultra Rapid Lispro Insulin (URLi) in patients using the MiniMed 780G hybrid closed-loop system. The outcome will be assessed from the data collected via the CareLink system throughout the intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel-Aviv Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petrovski G, Campbell J, Pasha M, Day E, Hussain K, Khalifa A, van den Heuvel T. Simplified Meal Announcement Versus Precise Carbohydrate Counting in Adolescents With Type 1 Diabetes Using the MiniMed 780G Advanced Hybrid Closed Loop System: A Randomized Controlled Trial Comparing Glucose Control. Diabetes Care. 2023 Mar 1;46(3):544-550. doi: 10.2337/dc22-1692. PMID 36598841
- [Background] Petrovski G, Campbell J, Pasha M, Hussain K, Khalifa A, Umer F, Almajaly D, Hamdar M, Heuvel TVD, Edd SN. Twelve-Month Follow-up from a Randomized Controlled Trial of Simplified Meal Announcement Versus Precise Carbohydrate Counting in Adolescents with Type 1 Diabetes Using the MiniMed 780G Advanced Hybrid Closed-Loop System. Diabetes Technol Ther. 2024 Mar;26(S3):76-83. doi: 10.1089/dia.2023.0429. PMID 38377327
- [Background] Warren M, Bode B, Cho JI, Liu R, Tobian J, Hardy T, Chigutsa F, Phillip M, Horowitz B, Ignaut D. Improved postprandial glucose control with ultra rapid lispro versus lispro with continuous subcutaneous insulin infusion in type 1 diabetes: PRONTO-Pump-2. Diabetes Obes Metab. 2021 Jul;23(7):1552-1561. doi: 10.1111/dom.14368. Epub 2021 Mar 23. PMID 33687783
- [Background] Datye KA, Boyle CT, Simmons J, Moore DJ, Jaser SS, Sheanon N, Kittelsrud JM, Woerner SE, Miller KM; T1D Exchange. Timing of Meal Insulin and Its Relation to Adherence to Therapy in Type 1 Diabetes. J Diabetes Sci Technol. 2018 Mar;12(2):349-355. doi: 10.1177/1932296817728525. Epub 2017 Sep 12. PMID 28895431
- [Background] Arrieta A, Battelino T, Scaramuzza AE, Da Silva J, Castaneda J, Cordero TL, Shin J, Cohen O. Comparison of MiniMed 780G system performance in users aged younger and older than 15 years: Evidence from 12 870 real-world users. Diabetes Obes Metab. 2022 Jul;24(7):1370-1379. doi: 10.1111/dom.14714. Epub 2022 May 12. PMID 35403792
- [Background] Bergenstal RM, Beck RW, Close KL, Grunberger G, Sacks DB, Kowalski A, Brown AS, Heinemann L, Aleppo G, Ryan DB, Riddlesworth TD, Cefalu WT. Glucose Management Indicator (GMI): A New Term for Estimating A1C From Continuous Glucose Monitoring. Diabetes Care. 2018 Nov;41(11):2275-2280. doi: 10.2337/dc18-1581. Epub 2018 Sep 17. PMID 30224348
- [Background] Choudhary P, Kolassa R, Keuthage W, Kroeger J, Thivolet C, Evans M, Re R, de Portu S, Vorrink L, Shin J, Habteab A, Castaneda J, da Silva J, Cohen O; ADAPT study Group. Advanced hybrid closed loop therapy versus conventional treatment in adults with type 1 diabetes (ADAPT): a randomised controlled study. Lancet Diabetes Endocrinol. 2022 Oct;10(10):720-731. doi: 10.1016/S2213-8587(22)00212-1. Epub 2022 Sep 1. PMID 36058207